CLINICAL TRIAL: NCT05391581
Title: The Role of the Intestinal Hormones Glucose-dependent Insulinotropic Polypeptide (GIP) and Glucagon-like Peptide 2 (GLP-2) in Postprandial Splanchnic Blood Flow Distribution and Metabolism in Humans
Brief Title: The Role of GIP and GLP-2 in Postprandial Splanchnic Blood Flow Distribution and Metabolism
Acronym: GA-17
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GA-17
Record Dates: First submitted 2022-05-06; First posted 2022-05-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Blood Flow
Keywords: Gut hormones; GIP; GLP-2; Physiology

STUDY DESIGN:
Intervention Model Description: Single blind, placebo controlled, randomized, crossover study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SAL-WAT (Placebo Comparator): Saline infusion, saline injection, water ingestion
  Interventions: Other: Placebo
- SAL-GLU (Active Comparator): Saline infusion, saline injection, glucose ingestion
  Interventions: Other: Placebo
- SAL-GIP (Active Comparator): Saline infusion, GIP injection, water ingestion
  Interventions: Other: Placebo
- SAL-GLP-2 (Active Comparator): Saline infusion, GLP-2 injection, water ingestion
  Interventions: Other: Placebo
- GIA-WAT (Experimental): GIPR antagonist infusion, saline injection, water ingestion
  Interventions: Other: GIPR antagonist / study tool; Other: Placebo
- GIA-GLU (Experimental): GIPR antagonist infusion, saline injection, glucose ingestion
  Interventions: Other: GIPR antagonist / study tool
- GLA-WAT (Experimental): GLP-2R antagonist infusion, saline injection, water ingestion
  Interventions: Other: GLP-2R antagonist / study tool; Other: Placebo
- GLA-GLU (Experimental): GLP-2R antagonist infusion, saline injection, glucose ingestion
  Interventions: Other: GLP-2R antagonist / study tool

INTERVENTIONS:
Other: GIPR antagonist / study tool — Selective antagonist of the GIPR, GIP(3-30)NH2
  Arms: GIA-GLU; GIA-WAT
Other: GLP-2R antagonist / study tool — Selective antagonist of the GLP-2R, GLP-2(3-33)
  Arms: GLA-GLU; GLA-WAT
Other: Placebo — Saline
  Arms: GIA-WAT; GLA-WAT; SAL-GIP; SAL-GLP-2; SAL-GLU; SAL-WAT

SUMMARY:
This project will describe the mechanisms of action and the relative contributions of GIP and GLP-2 to changes in gastrointestinal blood flow induced by oral glucose, exogenous GIP and GLP-2 infusions, and endogenous GIP and GLP-2 with the use of two novel receptor antagonists GIP(3-30)NH2 and GLP-2(3-33) in healthy individuals.

DETAILED DESCRIPTION:
Each participant will attend eight independent randomised experimental days in the MRI-scanner with intravenous infusion (hormone/placebo), subcutaneous injection (hormon/placebo) and oral ingestion (glucose/water). On experimental day A-C, an intravenous infusion of saline, GIP(3-30)NH2, or GLP-2(3-33), respectively, starts at time point -20 minutes. On experimental day D-F, the same infusions are combined with an oral glucose tolerance test (75 gram of glucose dissolved in 250 ml water ingested orally) at time point 0 minutes. On experimental days G-H, a subcutaneous injection of either GIP or GLP-2 at time point 0 minutes is performed (positive control) during saline infusion and oral water ingestion.

MRI measurements are repeatedly performed and blood samples are drawn to be analysed for endocrine responses from the intestines, pancreas, and bones.

ELIGIBILITY:
Inclusion Criteria:

* No first degree relatives with diabetes
* BMI 20-27 kg/m2

Exclusion Criteria:

* Not MRI-compatible implants
* Claustrophobia
* Diabetes
* Abnormal kidney or liver function
* Anemia
* Planned weight loss or change in diet
* Hypertension
* Other conditions that could be expected to affect the primary or secondary outcomes

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Redistribution of splanchnic blood flow (functional MRI) | 90 minutes
  Flow in mesenteric superior artery

SECONDARY OUTCOMES:
GIP levels | 90 minutes
  Blood sample (pmol/L)
GLP-2 levels | 90 minutes
  Blood sample (pmol/L)
GIP(3-30)NH2 levels | 90 minutes
  Blood sample (nmol/L)
GLP-2(1-33) levels | 90 minutes
  Blood sample (nmol/L)
CTX (bone resorption marker) | 90 minutes
  Blood sample
P1NP (bone formation marker) | 90 minutes
  Blood sample
Glucose | 90 minutes
  Blood sample (mmol/L)
C-peptide | 90 minutes
  Blood sample (pmol/L)
Insulin | 90 minutes
  Blood sample (pmol/L)
Glucagon | 90 minutes
  Blood sample (pmol/L)
Heart rate | 90 minutes
  Beats/minute
Flow in coeliac trunk | 90 minutes
  Functional MRI estimated blood flow
Flow in hepatic artery | 90 minutes
  Functional MRI estimated blood flow
Flow in portal vein | 90 minutes
  Functional MRI estimated blood flow
Liver oxygen content | 90 minutes
  Functional MRI estimated oxygenation

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Will share upon requests
Supporting Information: Study Protocol, CSR, Analytic Code